CLINICAL TRIAL: NCT05211830
Title: A Phase I/II, Multicenter, Randomized, Double-blind, Placebo Within-patient Controlled, First-in-human (FIH) Proof of Concept (PoC) Study to Evaluate the Safety and Efficacy of Topically Applied SXR1096 Cream in Patients With Netherton Syndrome (NS)
Brief Title: A Study to Evaluate Topically Applied SXR1096 Cream in Patients With Netherton Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sixera Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SXR001
Record Dates: First submitted 2021-10-14; First posted 2022-01-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will act as their own controls as they will all be treating different contralateral areas of the skin with active and placebo creams in a blinded fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and placebo will be provided in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SXR1096 cream (Experimental): The active treatment will be the specific small molecule inhibitor of KLK5, 7 and 14 in a proprietary skin cream formulation.
  Interventions: Drug: SXR1096 cream
- Placebo cream (Placebo Comparator): The placebo control will be the proprietary skin cream formulation without the active substance.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: SXR1096 cream — Skin cream to be applied twice a day to a predefined area of the skin
  Arms: SXR1096 cream
Drug: Placebo cream — Skin cream to be applied twice a day to a predefined area of the skin
  Arms: Placebo cream

SUMMARY:
In this phase I/II trial a topical skin cream with the active substance SXR1096 will be tested in patients with Netherton syndroms, a rare inflammatory skin disease. SXR1096 is a specific and potent protease inhibitor that can inhibit the proteases kallikrein 5, 7 and 14 - all recognised as up-regulated and causing the disease state in Netherton syndrome patients. Patients will be treated for one month with active cream and placebo cream at different areas of the skin.

DETAILED DESCRIPTION:
Netherton syndrome is a ultra-rare and very severe form of ichtyosis. It is a mongenetic disease. There is no specific treatment available for Netherton syndrome.

In this phase I/II trial a topical skin cream with the active substance SXR1096 will be tested in patients with Netherton syndrom. SXR1096 is a specific and potent protease inhibitor that can inhibit the proteases kallikrein 5, 7 and 14 - all recognised as up-regulated and causing the disease state in Netherton syndrome patients, as these patients have a gene defect in the gene spink5 encoding for the protease inhibitor LEKTI - that will normally regulate the activity of KLK5, 7 and 14 in the stratum corneum of the skin,

Patients will be treated for one month with active cream and placebo cream at different areas of the skin. The study will assess the safety and efficacy of the treatment in patients. There will also be pharmacokinetic, pharmacodynamic and biomarker studies conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years at the screening visit and also adolescents (12-17 years) only after initial cohort of 5 adult patients have been treated for at least three days.
2. Patients/legal guardian endpoint must be willing to provide written informed consent.
3. Clinical diagnosis of NS including at least 3 out of the 4 following clinical criteria;

   1. Neonatal erythroderma
   2. Bamboo hair and/or alopecia
   3. Chronic atopy specified as food allergy, asthma, rhino conjunctivitis and/or eczema for at least 2 years
   4. Ichthyosis linearis circumflexa
4. Patients must be willing and able to understand and can comply with study requirements, apply the medication as instructed and be able to complete the study.
5. Absent LEKTI on immunohistochemistry of skin biopsy and/or confirmed mutation in SPINK5 gene
6. NS involvement ≥ 20% of Body Surface Area (BSA) required at both the screening and baseline visits.
7. Investigator Global Assessment (IGA) of two areas to be treated, score ≥3, i.e. moderate or severe for each area required. Each target area approx. 9% of BSA. i.e. equal to one arm.
8. Female of childbearing potential must either commit true abstinence when this is in line with the preferred and usual lifestyle or use an adequate and approved method of contraception throughout the study and for 4 weeks after the last study drug application. This criterion also applies to a prepubertal female subject who begins menses during the study.

Adequate and approved methods of contraception applicable for the subject and/or her partner are defined below:

* Progestogen-only oral hormonal contraception
* Combination of male or female condom with cap, diaphragm, or sponge with spermicide (double barrier methods)
* Combined (estrogen- and progestogen-containing) oral, intravaginal, or transdermal hormonal contraception
* Injectable or implanted hormonal contraception
* Intrauterine devices or intrauterine hormone-releasing system
* Bilateral tubal ligation or tube insert (such as the Essure system) at least 3 months before the study
* Vasectomy of partner at least 3 months before the study
* Female subjects of non-childbearing potential must meet one of the following criteria:
* Absence of menstrual bleeding for 1 year prior to screening without any other medical reason
* Documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before screening

Exclusion Criteria:

1. Female patient who is pregnant, nursing an infant or planning a pregnancy throughout the course of the study
2. Patient with any uncontrolled systemic disease. A potential patient in whom therapy for a systemic disease is not yet stabile for at least 3 months will not be considered for entry into the study.
3. Patient with positive serology tests like HIV, HCV & HBsAg.
4. Patient with presence of any skin disease that might interfere with the diagnosis or evaluation of the test medications. Cutaneous infection within 1 week before the baseline visit or, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks before the baseline visit.
5. Patient that has a condition or is in a situation, which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.
6. Use of topical drugs that might alter the course of NS (e.g., topical corticosteroids and topical calcineurin inhibitors) within two weeks before baseline visit.
7. Patient with a known sensitivity to any of the study treatments and/or their components.
8. Patient who anticipates a need to use other topical or systemic therapy that might alter the course of NS. Emollients/creams can be used on remaining skin area but not the test areas. Use of topical prescription treatment within 2 weeks prior to initial dosing of study drug. Recent systemic treatment for NS (e.g. systemic corticosteroids, antibiotics, immunosuppressant, biologic and biosimilars treatments). A washout period of 4 weeks will be required for such patients to be eligible to participate in the trial.
9. Patient who anticipates the need for surgery or hospitalization during the study.
10. Concurrent involvement in any other clinical study/expanded access program with an investigational drug or device, or participation in a clinical study within 30 days prior to entering the study.
11. Suspected or confirmed COVID-19 infection within 4 weeks before the screening or baseline visit. Unresolved COVID-19 infection. Planned vaccination for COVID-19 during screening, treatment period or before the follow-up visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Safety of the treatment with SXR1096 compared to placebo in initial cohort of adults | 4 week
  Number of patients with treatment-related adverse events during the treatment period of 4 weeks
Safety of the treatment with SXR1096 compared to placebo in adults and adolescents | 4 weeks
  Number of patients with treatment-related adverse events during the treatment period of 4 weeks
Efficacy of the treatment with SXR1096 compared to placebo in adults and adolescents | 4 weeks
  The change in Investigator Global Assessment (IGA) score 0-4 at EOT compared to baseline (0 being clear of lesions (erythema and scaling) and 4 being the worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Maarten de Chateau, MD PhD, Study Director — Sixera Pharma
Locations (5):
- Medical University Innsbruck, Tirol Kliniken, Innsbruck, Austria
- France (2):
  - Saint Louis Hospital, Paris
  - Necker Hospital, Paris
- University of Freiburg, Freiburg im Breisgau, Germany
- Karolinska Hospital, Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No